CLINICAL TRIAL: NCT01468480
Title: Comparison of Human Pulpal Response After Pulpal Exposure to Common Treatments and Single-visit MTA
Brief Title: Human Pulpal Response After Pulp Capping With Four Different Agents
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Mahta Fazlyab, Post graduate student of endodontics, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: p/261/d
Record Dates: First submitted 2011-11-04; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Dental Pulp Exposure
Keywords: direct pulp capping; MTA; Single visit pulp cap; Multical
MeSH Terms: conditions — Dental Pulp Exposure | interventions — mineral trioxide aggregate; Dycal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pro Root MTA- standard method (Experimental): application of MTA in second group and 24 hour interval before restoration
  Interventions: Drug: Pro Root MTA
- Pro Root MTA- single visit (Experimental): Intervention/Control application of MTA in third group and 15 minute interval before restoration
  Interventions: Drug: Pro Root MTA- single visit
- MultiCal / LimeLite (Experimental): application of Multical in forth group
  Interventions: Drug: MultiCal
- Dycal (Active Comparator): application of Dycal in first group as a pulp dressing agent
  Interventions: Drug: Dycal

INTERVENTIONS:
Drug: Pro Root MTA — application of MTA in second group and 24 hour interval before restoration
  Other Names: Mineral Trioxide Aggregate
  Arms: Pro Root MTA- standard method
Drug: Pro Root MTA- single visit — application of MTA in third group and 15 minute interval before restoration
  Other Names: Mineral Trioxide Aggregate
  Arms: Pro Root MTA- single visit
Drug: MultiCal — application of Multical in forth group as a pulp dressing agent
  Other Names: Hard set calcium hydroxide paste
  Arms: MultiCal / LimeLite
Drug: Dycal — application of Dycal in first group as a pulp dressing agent
  Other Names: chemical set calcium hydroxide
  Arms: Dycal

SUMMARY:
Application of four different pulp capping methods on human sound premolars after intentional exposure of the buccal pulp horn through a class one occlusal cavity.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to compare the effect of different direct pulp capping methods on human pulpal response in the terms of inflammation & dentinal bridge formation. Methods: Eight patients providing 32 sound first premolars are selected. As recommended by ISO / TC 7405 pulpal exposure will be performed through a class I cavity. Four groups of eight specimens each will be defined according to the pulp capping method. Group A, will receive chemical set calcium hydroxide (Dycal). Group B, will receive mineral Trioxide Aggregate (MTA) according to manufacturer's instruction. Group C, will receive MTA and after its primary setting, within 15 minutes, the cavity is restored in the same appointment. Group D, will receive Multical as a direct pulp capping agent. Specimens will be assessed in the terms of dentinal bridge formation, its appearance compared to natural dentin, its thickness and inflammatory pulpal response. The last item will be scored 0-3 in which 0 corresponds to none, 1 to minimal, 2 to moderate and 3 to severe inflammation. In case of an abscess or true tissue necrosis, a score of 4 will be given as recommended by ISO / TC 7405.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging from 10 to 16
* Patients who need to extract 4 premolars for orthodontic purposes
* the teeth should be free of caries and clinical symptoms
* Through thermal tests and radiographic examination absence of any pathology is confirmed.
* Periapical radiographs demonstrating absence of any pathology
* no sensitivity to percussion, palpation and biting, no sensitivity to cold after 5 seconds contact with Green Endo Ice refrigerant spray, heat sensitivity after applying tempered Gutta Percha for 10 seconds.
* Absence of any systematic disorder
* No consumption of drugs of any kind
* All patients and their parents need to sign a fully informed consent.

Exclusion Criteria:

* If any of the teeth shows caries, restoration, crack or hypocalcification
* presence of any periapical pathosis
* Teeth that seem sensitive to cold, hot, percussion or pressure
* any systematic disorder
* consumption of drugs of any kind.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2010-06; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
histologic findings - inflammation of the pulp | 6weeks
  According to histological evaluation and ISO/DIS7405, the investigators gave to non inflamed cases no points, mild cases 1 point, moderate cases 2 points, severe cases 3 points and necrosis 4 points.

SECONDARY OUTCOMES:
histologic findings - formation of the dentinal bridge | 6 weeks
  The specimens will be evaluated in the terms of dentinal bridge formation and its resemblence to natural dentin and also the thickness of the bridge.

CONTACTS AND LOCATIONS:
Overall Officials: Mahta Fazlyab, Resident, Principal Investigator — Fazlyab Mahta
Locations (1):
- Mahta Fazlyab, Tehran, Tehran Province, Iran